CLINICAL TRIAL: NCT02386124
Title: Frailty Assessment in eldeRly Admitted to hoSpital for acutE caRdiac Disease Prospective Study
Brief Title: Frailty in Elderly Patients Receiving Cardiac Interventional Procedures
Acronym: FRASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, MD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140994
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Aged
Keywords: frailty; elderly; acute coronary syndrome; acute heart failure; arrhythmias
MeSH Terms: conditions — Frailty; Acute Coronary Syndrome; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- frailty evaluation (Other): all consecutive patients admitted to hospital for acute cardiac disease aged more than 69 years will be evaluated with Short Portable Mental Status Questionnaire (SPMSQ), handgrip and Short Physical Performance Battery (SPPB).
  These three tests (SPMSQ, SPPB and handgrip) are the intervention of the study. They are the assays to establish the frailty status
  Interventions: Other: frailty evaluation

INTERVENTIONS:
Other: frailty evaluation — assessment of mental and physical frailty before discharge from cardiac departement

SUMMARY:
In Italy, life expectancy at birth has reached 80 years in men and 85 in women; in about 50 years, life expectancy at the age of 80 has increased by an extraordinary 61% and 55%, respectively, due to more effective therapies and lower mortality of many diseases. Yet, chronic diseases are nowadays more important, and often coexist as comorbidity or multimorbidity, depending on whether an index condition has been considered. These conditions increase the risk of death and reduce functional autonomy in the elderly and, therefore, should be carefully considered within comprehensive geriatric assessment. The epidemiology of cardiovascular disease, as demonstrated among others by the Oxford Vascular Study, shows a clear trend in age-dependent, as the number of events and their incidence increases with age, and about half are concentrates over 75 years.

In addition, some observational studies in elderly patients have suggested an association between frailty and cardiovascular disease: fragility and cardiovascular disease share a common biological pathway, and cardiovascular diseases may accelerate the onset of frailty. The frailty syndrome was identified in 25% to 50% of patients with cardiovascular disease, according to the rating scale used and the population studied. Frail patients with cardiovascular disease, in particular those undergoing invasive procedures or suffering from coronary artery disease and aortic valve disease, have a much higher adverse events and complications, suggesting the need for a more accurate functional stratification and a more careful evaluation of the risk/benefit ratio of some invasive procedures.

Among the numerous tests proposed in the literature for the functional evaluation and objective measures of physical capability in elderly patient, the Short Physical Performance Battery (SPPB) and the evaluation of hand grip strength (grip strength) are those characterized by an improved prognostic ability and an easy administration.

The present study is performed to assess if SPPB and handgrip are helpful to better stratify the prognosis (all-causes death and hospital admission for all causes) in elderly patients admitted to hospital for cardiac causes.

DETAILED DESCRIPTION:
This is a prospective observational study. This a multicenter study involving 4 Italian Cardiology Units (Ferrara, Cento, Forlì, Ravenna).

The study is expected to enroll at least 400 consecutive patients with ≥70 years, which are admitted to our cardiovascular departement for:

* GROUP A: acute coronary syndrome,
* GROUP B: bradycardia or tachyarrhythmias requiring device implantation (pace-maker, implantable cardioverter defibrillator, cardiac resynchronization therapy)
* GROUP C: acute heart failure.
* GROUP D: symptomatic severe aortic stenosis receiving aortic valve replacement or aortic balloon valvuloplasty or transcatheter aortic valve implantation.

The main group of the study is the group A. The Authors will enroll at least 300 patients of the group A. The main finding of the study will be for ACS patients. The results of group A will be reported by Authors in a separate and principal paper.

To generate hypothesis for future studies, the Authors will enroll also other groups of patients admitted to hospital for cardiac cause (group B, C and D). These patients will be object of separate publications.

In all patients, the following functional assessments will be performed before the hospital discharge:

* handgrip test (see definition below).
* Short Portable Mental Status Questionnaire (SPMSQ, see definition below).
* Short Physical Performance Battery (SPPB, see definition below).
* Multidimensional Prognostic Index (MPI, see definition below).

The aim of the study is to evaluate if SPPB value is able to stratify prognosis in elderly patients admitted to hospital for cardiac causes.

DEFINITION OF ACUTE CORONARY SYNDROME.

As suggested by current guidelines, we define a patient suffering from ACS if he meets the following criteria (the first mandatory which must add up to at least one criterion 2 or 3):

1. chest pain suggestive of cardiac origin lasting at least 20 minutes.
2. ECG changes compatible with signs of myocardial ischemia (ST over at least one mm in at least two contiguous leads or new onset left bundle branch block not known before or ST-segment depression of at least one mm in at least two contiguous leads or negative/ flattening of T wave)
3. detection of rise of cardiac biomarker values with at least one value above the 99th percentile of the upper reference in two consecutive blood samples

DEFINITION OF ACUTE MYOCARDIAL INFARCTION (ESC GUIDELINES 2012)

The term acute myocardial infarction should be used in case of evidence of myocardial necrosis in a clinical picture compatible with acute myocardial ischemia. And in particular it must verify detection of movement enzyme preferentially typical of troponin above the 99th percentile than the limit of the standard and in the presence of at least one of the following conditions:

* Symptoms of ischemia,
* Changes in de novo ST-segment and T-wave, new-onset left bundle branch block, development of pathological Q waves on the ECG.
* Evidence of loss of viable myocardium imaging or detection of new wall motion defects,
* Identification of an intracoronary thrombus on coronary angiography.

DEFINITION OF HEART FAILURE (ESC GUIDELINES 2012) It defines heart failure or an abnormality of the structure of the cardiac function that involves an insufficient ability of the heart to provide for the oxygen requirements in relation to the metabolic demands of the tissues, despite normal or increased filling pressures. Heart failure is a syndrome that is characterized by the presence of typical symptoms (dyspnea, peripheral edema and fatigue) and signs resulting from an abnormality of cardiac structure and function.

DEFINITION AND METHODS OF ASSESSMENT TEST DELL'HANDGRIP (HGT). The handgrip test measures the force of contraction of the flexor muscles of the fingers through the use of a dynamometer. From literature it is known as such index correlates with the eventual malnutrition of the subject, with its capacity of recovery and functional recovery post-surgery, as well as to be in relation with age. The measurement will be made at the time of admission, namely within 24 hours of admission in acute coronary care in the event that the patient is admitted with a diagnosis of acute myocardial infarction with ST-segment elevation or before being subjected to coronary angiography in case aortic valve disease or acute coronary syndrome without ST-segment elevation, under the supervision and assistance of medical staff. In each patient, three measurements will be carried out. Will be taken into consideration for the study the highest value. The measurement will be performed as indicated by current guidelines, with the patient seated, with the dominant hand and the elbow flexed 90°. They are well known limitations of the method and its variability. At the same time this method was chosen because it is not laborious, virtually cost-free, well-administered in all patients admitted for ACS or aortic valve disease and therefore readily identifiable as a method of coarse screening in elderly patients without known diagnosis of "frail elderly" but at risk to be. All medical personnel involved in the study performed a specific course to learn the proper management and execution of screening with handgrip tes and has personal experience in its proper execution.

SHORT PHYSICAL PERFORMANCE BATTERY (SPPB). The scale SPPB is a short battery of tests created to evaluate the functionality of the lower limbs. This battery is made up of 3 different sections designed to assess a balance with 3 tests: the maintenance of the position with the feet together for 10 seconds then the semi-tandem and finally tandem again for 10 seconds. The score of this section varies from a minimum of 0 if the patient is unable to maintain position with your feet together for at least 10 seconds to a maximum of 4 if he can accomplish all three tests. The second section of the test is intended to evaluate the progress of 4 linear meters and depending on the time of the performance section of the score ranges from 0 if unable, at one point if the performance has a longer duration of 8.7 seconds, for a up to 4 if he can accomplish the task in less than 4.80 sec. The third section investigates the ability of the battery to run for 5 consecutive times, getting up from a chair without using the arms in this regard that must be crossed in front of chest. Also in this case, the score ranges from 0 incapable or if the performance has a duration greater than 60 seconds, to a maximum of 4 if such performance is carried out in less than 11.20 seconds. The scores range from 0 (worst performance) to 12 (best performance).

A score between 5 and 9 shows seniors still independent, but with reduced physical performance, which can therefore be regarded as fragile and high risk, deserving of special attention and specific interventions, acts to reduce the risk of adverse consequences. Data in the literature confirm that the SPPB correlates with the risk of developing disability in BADL and mobility, in proportion to the decrease of the SPPB score, regardless of age, sex and presence of certain chronic diseases. The SPPB score then emerges as a powerful predictor of disability and mortality in the elderly population. The battery SPPB proved to be a valid predictor of prognosis in heart patients: in elderly hospitalized for acute exacerbation of chronic heart failure, the SPPB score at discharge was able to predict the long-term mortality. This assessment thus appears to be safe and feasible in hospitalized patients: test will be performed in patients with hemodynamic stabilization prior to discharge.

MULTIDIMENSIONAL PROGNOSITC INDEX (MPI)

The Multidimensional Prognostic Index (MPI) is a prognostic tool based on a standard Comprehensive Geriatric Assessment (CGA) that predicts short- and long-term mortality in elderly subjects. The MPI includes 63 items distributed in 8 domains of CGA as follows:

1. Activities of Daily Living (ADL): 6 items
2. Instrumental Activities of Daily Living (IADL): 8 items
3. Short Portable Mental Status Questionnaire (SPMSQ): 10 items
4. Mini Nutritional Assessement (MNA): 18 items
5. Exton-Smith Scale (ESS): 5 items
6. Cumulative Index Rating Scale - Comorbidity Index (CIRS-CI): 14 items
7. Number of drugs used: 1 item
8. Co-habitation status: 1 item On the basis of MPI values, it is possible to calculate the short- and long-term mortality risk of the older subjects and to define the severity grade of mortality risk: low, moderate and severe. Several studies showed that the prognostic accuracy of the aggregated MPI was significantly greater than the prognostic accuracy of its individual components considered singularly. Thus the multidimensional approach can be successfully used in elderly patients for both clinical and administrative purposes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥70
* hospital admission in the cardiac department for acute cardiac disease (acute coronary syndromes, acute heart failure, arrhythmias requiring pace-maker or implantable cardioverter-defibrillator)

Exclusion Criteria:

* SPMSQ value ≤4
* inability to stay upright
* life expectancy <3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 402 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
composite endpoint of all-cause mortality and all-cause hospital admission | 1 year
  1-year cumulative incidence of all-cause mortality and all-cause hospital admission

SECONDARY OUTCOMES:
all-cause mortality | 1 year
  1-year cumulative incidence of death for all-causes
hospital admission for all-causes | 1 year
  1-year cumulative incidence of hospital admission for all causes
cardiac adverse events | 1 year
  1-year cumulative incidence of cardiac death, myocardial infarction, heart failure

OTHER OUTCOMES:
cerebrovascular accident | 1 year
  1-year cumulative incidence of stroke and/or transient ischemic attack
admission in emergency room | 1 year
  1-year cumulative incidence of admission in emergency room
arrhythmias | 1 year
  1-year cumulative incidence of new diagnosis of significant arrhythmias
severe aortic stenosis | 1 year
  1-year cumulative incidence of new diagnosis of severe aortic stenosis
acute coronary syndrome (ACS) | 1 year
  1-year cumulative incidence of new diagnosis of ACS (unstable angina and myocardial infarction)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Campo, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara; Stefano Volpato, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Campo G, Pavasini R, Maietti E, Tonet E, Cimaglia P, Scillitani G, Bugani G, Serenelli M, Zaraket F, Balla C, Trevisan F, Biscaglia S, Sassone B, Galvani M, Ferrari R, Volpato S. The frailty in elderly patients receiving cardiac interventional procedures (FRASER) program: rational and design of a multicenter prospective study. Aging Clin Exp Res. 2017 Oct;29(5):895-903. doi: 10.1007/s40520-016-0662-y. Epub 2016 Oct 28. PMID 27796963
- [Derived] Balla C, Passarini G, Bonsi B, Pavasini R, Tonet E, Malagu M, Campo G, Bertini M. Physical performance status predicts mortality in aging patients undergoing pacemaker implantation. J Cardiovasc Med (Hagerstown). 2021 Oct 1;22(10):738-743. doi: 10.2459/JCM.0000000000001209. PMID 33973534
- [Derived] Pavasini R, Maietti E, Tonet E, Bugani G, Tebaldi M, Biscaglia S, Cimaglia P, Serenelli M, Ruggiero R, Vitali F, Galvani M, Minarelli M, Rubboli A, Bernucci D, Volpato S, Campo G. Bleeding Risk Scores and Scales of Frailty for the Prediction of Haemorrhagic Events in Older Adults with Acute Coronary Syndrome: Insights from the FRASER study. Cardiovasc Drugs Ther. 2019 Oct;33(5):523-532. doi: 10.1007/s10557-019-06911-y. PMID 31549262
- [Derived] Campo G, Maietti E, Tonet E, Biscaglia S, Ariza-Sole A, Pavasini R, Tebaldi M, Cimaglia P, Bugani G, Serenelli M, Ruggiero R, Vitali F, Formiga F, Sanchis J, Galvani M, Minarelli M, Lucchi GR, Ferrari R, Guralnik J, Volpato S. The Assessment of Scales of Frailty and Physical Performance Improves Prediction of Major Adverse Cardiac Events in Older Adults with Acute Coronary Syndrome. J Gerontol A Biol Sci Med Sci. 2020 May 22;75(6):1113-1119. doi: 10.1093/gerona/glz123. PMID 31075167